CLINICAL TRIAL: NCT06600880
Title: Neuronavigation-guided Focused Ultrasound-induced Blood-brain Barrier Opening in Alzheimer's Disease Patients and Its Effects on Brain Amyloid and Tau
Brief Title: Neuronavigation-guided FUS-induced BBB Opening in Alzheimer's Disease Patients and Its Effects on Brain Amyloid and Tau
Acronym: FUS-AD
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: AAAV4854
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — Magnetic Resonance Spectroscopy; florbetapir; MK-6240; gadoterate meglumine; Blood Specimen Collection; Urinalysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Focused ultrasound treatment (Experimental): Neuronavigation-guided focused ultrasound treatment in Alzheimer's disease patients using a single-element transducer in conjunction with microbubbles.
  Interventions: Device: Neuronavigation-guided single-element focused ultrasound transducer; Drug: Lumason; Other: Magnetic Resonance Imaging (MRI) with or without gadolinium contrast agents; Radiation: Positron Emission Tomography (PET); Drug: Amyvid; Drug: MK-6240; Drug: Dotarem; Diagnostic Test: Blood draw; Device: UR5e; Diagnostic Test: Urine test

INTERVENTIONS:
Device: Neuronavigation-guided single-element focused ultrasound transducer — Non-invasive focused ultrasound-induced blood-brain barrier opening will be attempted using a single-element transducer, guided with a neuronavigation system.
Drug: Lumason — New packages of Lumason microbubbles will be shipped from Bracco Diagnostics Inc. and will be used in conjunction with the ultrasound transducer to temporarily open the BBB. Lumason microbubbles will be freshly activated before treatment sonication and will be drawn using a 10-ml syringe to reach the desired dosage of 0.1mL/kg right before the intravenous injection.
Other: Magnetic Resonance Imaging (MRI) with or without gadolinium contrast agents — A high-resolution MRI (with and without gadolinium (Dotarem) contrast agent) will be acquired prior to BBB opening on the GE SIGNATM Premier (3T) (same scanner as in the NHP study) for pre-treatment planning and screening purposes. Then, a second MRI (with and without gadolinium) will be acquired and read by a Board-Certified Radiologist immediately after the treatment sonication in order to assess the BBB opening and safety. Finally, a final follow-up MRI (with and without gadolinium) will be conducted 3 days (±1 day) after the treatment to confirm BBB closing and/or safety. This will be read by a Board-Certified Radiologist as well.
  All MRI procedures will be performed at the CUIMC/Neurological Institute of New York.
Radiation: Positron Emission Tomography (PET) — A first PET/CT scan with Amyvid (18F-Florbetapir) and MK-6240 (F18-Florquinitau) tracers will be performed on the SIEMENS Biograph 64 to assess the baseline amyloid plaque load and tau load before the treatment, respectively. Finally, two follow-up PET/CT scans will be conducted 3 weeks (±1 week) and 3 months (±2 weeks) post-treatment to assess amyloid plaque load (using Amyvid) and tau load (using MK-6240).
Drug: Amyvid — Amyloid PET tracer Amyvid (18F- Florbetapir) will be stored in their original container with proper radiation shielding at 25 °C and only handled by properly trained personnel in the handling and administration of radioactive materials, which requires employing proper radiation protection procedures.
  Other Names: 18F-Florbetapir
Drug: MK-6240 — [18F]MK-6240 will be synthesized, purified, and formulated at the local radiochemistry synthesis laboratory and will be administered as a sterile, pyrogen-free solution by IV injection. The radiotracer [18F]MK-6240 is supplied in a sterile, ready-to-use solution, direct from the Columbia University PET Center. It is supplied for a targeted calibration time, the precise volume to be administered at a given time can be calculated based on the decay of F-18. Only personnel properly trained in the handling and administration of radioactive materials should handle [18F]MK-6240. Usual radiation protection procedures should be used for handling radiotracers, including shielding (lead or tungsten containers/shields), and personal protective equipment including gloves. There are no specific procedures required for the handling of [18F]MK-6240. The expiry of [18F]MK-6240 is eight hours from the time at End of Synthesis (EOS).
Drug: Dotarem — FDA-approved medication. Dotarem will be handled in accordance with the CUMC Research Pharmacy procedures and NYP policy P168, Version 4. Dotarem will be used according to its labeling. 0.2 ml/kg.
Diagnostic Test: Blood draw — Blood samples will be collected through an intravenous catheter or a finger prick during screening, on the day of the FUS treatment and the follow up examinations (week 3 and month 3). These samples will be processed to assess any blood content changes induced by the focused ultrasound treatment.
Device: UR5e — Universal Robots robotic arm used for the accurate positioning of the neuronavigation-guided single-element focused ultrasound transducer with respect to the patient's head.
Diagnostic Test: Urine test — Urine test required following the MRI and PET Centers policy used clinically for pregnancy screening

SUMMARY:
The primary purpose of this phase 1b study is to further assess the safety and reversibility of focused ultrasound induced blood-brain barrier opening (FUS-BBBO) in participants with Alzheimer´s Disease (AD) using a single-element transducer with neuronavigation guidance. Preliminary results from our phase 1a study demonstrate that our neuronavigation-guided FUS system was capable of safely and transiently open the BBB in participants with AD. The information collected in this new study may be used to design future clinical trials to ultimately provide a viable alternative for treatment of AD in a safe and noninvasive manner.

Our secondary objective includes the assessment of the therapeutic efficacy of FUS-BBBO in reducing amyloid beta and neurofibrillary tangles, the main hallmark pathologies of AD, using PET tracers. Based on our preclinical studies in AD transgenic mouse models, FUS-BBBO alone was able to reduce both the amyloid beta and tau protein load, resulting in improvements in behavioral tasks assessing memory. Therefore, in this new study, the effect of FUS-BBBO on the amyloid beta and tau protein load in patients with AD will be assessed through the use of PET tracers.

DETAILED DESCRIPTION:
Regarding the primary purpose of this study, the human module for the neuronavigator was implemented in our phase 1a trial, and initial feasibility and safety in a small cohort of AD patients had been tested, with a fast procedural time that required no anesthesia.

Regarding the secondary objective, both amyloid beta and tau protein load in the brain will be assessed at baseline (before FUS-BBBO treatment), and 3-weeks and 3-months after FUS-BBBO treatment, to assess any short-term or long-term changes, respectively.

ELIGIBILITY:
Inclusion Criteria. AD patients will be recruited in person and have to be over 50 years of age and able to give consent. Patients diagnosed with MCI or AD will be included in our study. Other more severe symptomatic patients will be eligible to enroll, as long as they have the ability to consent for their participation. Screening is essential and will be performed by our collaborator and neurologist of the study, Dr. Lawrence Honig, MD at the Taub Institute of Alzheimer's Disease and Aging at Columbia. After the initial screening we will acquire MRI scans as part of the study and finalize enrollment or exclusion of the patient. Inclusion criteria thus include:

* Age greater than 50 years old.
* Diagnosis of MCI or AD. All following criteria must be met:
* MMSE score between 12 and 26.
* Modified Hachinski Ischemia Scale (MHIS) score of <= 4
* Short form Geriatric Depression Scale (GDS) score of <= 6.
* PET scan confirming amyloid plaque load using Amyvid (18F-Florbetapir).
* PET scan confirming tau positivity in the frontal lobe using MK-6240 (F18-Florquinitau).
* Ability to provide informed consent.

Exclusion Criteria. Exclusion criteria include surgeries and other pathologies not associated with AD, as outlined in the following list:

* Prior administration of any amyloid-reducing agent such as aducanumab or lecanemab.
* Contraindication for MRI.
* Contra-indication history or hypersensitivity to MRI contrast agents (e.g., Dotarem) or microbubbles (e.g., Definity, Lumason), including polyethylene glycol (PEG) allergy.
* Prior brain surgery, including deep brain stimulation.
* Metallic implants.
* Abnormal coagulation profile (significant abnormality in PT, PTT, or platelets).
* Anticoagulant therapy.
* History of seizure disorder.
* Brain atrophy to a degree that would interfere with ultrasound delivery.
* Inability to comply with the procedures of the protocol, including follow-up scans.
* Women with capacity to bear children or lactating.
* Impaired renal function with estimated glomerular filtration rate (eGFR) <30 mL/min/1.73m2 provided by a standard blood test 2-4 weeks prior to the ultrasound treatment.
* Active infection/inflammation.
* Acute or chronic hemorrhages, i.e. > 4 lobar microbleeds, or an area of siderosis or macrohemorrhages.
* Tumors or space-occupying lesions of significance.
* Any uncontrolled medical disorder that might interfere with the ability to safely perform the study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2026-08 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Total Number of Individuals With Successful Opening of the BBB | 4 days, including the day of treatment
  Opening the BBB successfully in all the patients, while obtaining a volume of BBB opened being similar and consistent for all patients

SECONDARY OUTCOMES:
Total Number of Safety Events Related to Opening of BBB | 4 days, including the day of treatment
  Showing safe BBB opening for all patients without any Adverse Event nor Serious Adverse Event, and showing its safety as well in 3 days after treatment
Percent Change in Amyloid PET Signal Intensity | 3 months (±2 weeks)
  A moderately shown in our previous clinical trial study, we expect to observe a slowed down increase of Amyloid protein load after the treatment on the two follow-ups performed at 3 weeks (±1 week) and 3 months (±2 week) after treatment.
Percent Change in MK-6240 PET Signal Intensity | 3 months (±2 weeks)
  As shown in our previous studies in mice, we expect to observe a slowed down increase or reduction on Tau protein load after the treatment on the two follow-ups performed at 3 weeks (±1 week) and 3 months (±2 week) after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Grace McIlvain, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
No individual participant data (IPD) will be shared with other researchers.